CLINICAL TRIAL: NCT01768013
Title: The Pharmacokinetics of LEO 90105 (Calcipotriol Hydrate Plus Betamethasone Dipropionate) in Japanese Subjects With Extensive Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCB 0904
Record Dates: First submitted 2013-01-10; First posted 2013-01-15 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2015-05

CONDITIONS: Psoriasis Vulgaris

ARMS (1):
- LEO 90105 Ointment (Experimental)
  Interventions: Drug: LEO 90105

INTERVENTIONS:
Drug: LEO 90105 — Once daily for four weeks

SUMMARY:
The pharmacokinetics of LEO 90105 (calcipotriol hydrate plus betamethasone dipropionate) in Japanese subjects with extensive psoriasis vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Japanese subjects having understood and signed a written informed consent form prior to any study related procedures being carried out (including activities related to the wash out period)
* 20 years of age or above.
* Either sex.
* Clinical diagnosis of psoriasis vulgaris amenable to topical treatment involving arms and/or trunk and/or legs.
* Psoriasis vulgaris on the trunk/limbs (excluding psoriasis on the genitals/skin folds) of not more than 30% body surface area (BSA)
* An Investigator's global assessment of disease severity (IGA) on area(s) to be treated of moderate, severe or very severe and a m-PASI score of ≥12.
* Females of childbearing potential must have a negative result for a urine pregnancy test at Day 1 (Visit 1) and must agree to use an adequate method of birth control, as judged by the (sub)investigator, during the study. The contraceptive method should have started an adequate amount of time before the pregnancy test, which is dependent on the particular method used and as judged by the (sub)investigator, and must continue for at least 1 week after the last application of study medication. A female is defined as not of child-bearing potential if she is postmenopausal (12 months with no menses without an alter-native medical cause) or surgically sterile (tubal ligation /section, hysterectomy or bilateral ovariectomy).

Exclusion Criteria:

* Systemic use of biological treatments with a potential effect on psoriasis vulgaris within the following time periods prior to Visit 1:
* etanercept, adalimumab, infliximab -3 months.
* ustekinumab - 4 months
* other products - within 3 months/5 half-lives (whichever is longer).
* Systemic treatments with all therapies other than biological treatments with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D analogues, retinoids, immu-nosuppressants such as ciclosporin and methotrexate) within 4 weeks prior to Visit 1 (use of inhaled and nasal corticosteroids is allowed, use of systemic antihistamines is allowed).
* Topical treatment of scalp psoriasis with vitamin D analogues (e.g. calcipotriol, tacalcitol, maxacalcitol), or very potent WHO group IV corticosteroids within 2 weeks prior to Visit 1.
* PUVA therapy, UVB therapy or UVA therapy within 4 weeks prior to Visit 1.
* Topical treatment of psoriasis on the face, genitals or skin folds with vitamin D analogues (e.g. calcipotriol, tacalcitol, maxacalcitol), or potent or very potent WHO group III or IV corticosteroids within 2 weeks prior to Visit 1.
* Topical treatment of psoriasis on area(s) to be treated with study medication within the 2-week period prior to Visit 1. (Use of emollients is allowed during this 2- week period, but not during the study.)
* Planned initiation of, or changes in, concomitant medication that may affect psoriasis vulgaris (e.g., beta-blockers, antimalaria drugs, lithium and ACE inhibitors) during the study.
* Topical treatment of conditions other than psoriasis with vitamin D analogues (e.g. calcipotriol, tacalcitol, maxacalcitol), or potent or very potent WHO group III or IV corti-costeroids within 2 weeks prior to Visit 1.
* Current diagnosis of erythrodermic, exfoliative, guttate or pustular psoriasis.
* Clinical signs or symptoms of Cushing's disease or Addison's disease
* Patients with any of the following disorders (a) or symptoms (b) present on the area(s) to be treated with study medication: (a) viral (e.g., herpes or varicella) lesions of the skin, fungal or bacterial skin infections, parasitic infections, skin manifestations in relation to syphilis or tuberculosis, rosacea, acne vulgaris, atrophic skin, striae atrophicae, ichthyosis, acne rosacea, ulcers, burns, frostbite, wounds, or (b) fragility of skin veins.
* Other inflammatory skin diseases (e.g., seborrhoeic dermatitis, contact dermatitis and cutaneous mycosis) that may confound the evaluation of psoriasis vulgaris.
* Planned excessive exposure of treated areas(s) to either natural or artificial sunlight (including tanning boths, sun lamps, etc) during the study.
* Known or suspected disorders of calcium metabolism associated with hypercalcaemia (subjects with results for albumin-corrected serum calcium above the reference range from the sample taken at the Washout/Screening Visit.
* Severe renal insufficiency, severe hepatic disorders or severe heart disease.
* Known or suspected hypersensitivity to components of the investigational products.
* Current participation in any other interventional clinical study
* Subjects who have received treatment with any non-marketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within the 4-week period prior to Visit 1 or longer, if the class of substance re-quires a longer washout as defined above (e.g. biological treatments).
* Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding
* Patients suspected of being unable to comply with the study protocol, e.g. due to alcoholism, drug dependence or psychotic state.
* Previous enrollment in this study.
* Hospitalised patients.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials at LEO Pharma — https://www.leopharmatrials.com/en

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject first visit: 09-Jul-2012 Last subject last visit: 30-Oct-2012
Pre-assignment Details: Prior to treatment at Visit 1, a washout period was completed if the subject was treated or had recently been treated with anti-psoriatic treatments or other relevant medication, as defined by the exclusion criteria. The washout period could last up to a maximum of 4 weeks.
Groups:
- LEO 90105 Ointment: Subjects received once daily topical treatment with LEO 90105 (calcipotriol hydrate plus betamethasone dipropionate ointment) on all lesions on the trunk and/or limbs (excluding psoriasis on the genitals and skin folds) for 4 weeks. Subjects were supplied with an amount of medication at day 1, day 7 and day 14 such that the maximum usage of LEO 90105 could be 90 g per week.
Period: Overall Study
Arm/Group | LEO 90105 Ointment
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  Japan | 13

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic: Cmax of Betamethasone Dipropionate
Description: The mean Cmax(Maximum Observed Plasma Concentration) of betamethasone dipropionate was determined.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

2. Primary Outcome: Pharmacokinetic: Cmax of Betamethasone Dipropionate
Description: The mean Cmax (Maximum Observed Plasma Concentration) of betamethasone dipropionate was determined
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

3. Primary Outcome: Pharmacokinetic: Cmax of Betamethasone Dipropionate
Description: The mean Cmax (Maximum Observed Plasma Concentration) of betamethasone dipropionate was determined
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

4. Primary Outcome: Pharmacokinetic: AUClast of Betamethasone Dipropionate
Description: The mean AUClast (Area under the Plasma Concentration-Time Curve from Time 0 to the Last Observed Measurable Concentration) for betamethasone dipropionate was determined
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

5. Primary Outcome: Pharmacokinetic: AUClast of Betamethasone Dipropionate
Description: as for outcome 4
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

6. Primary Outcome: Pharmacokinetic: AUClast of Betamethasone Dipropionate
Description: as for outcome 4
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

7. Primary Outcome: Pharmacokinetic: Cmax of Betamethasone 17-propionate
Description: The mean Cmax(Maximum Observed Plasma Concentration) of betamethasone 17- propionate was determined
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | 218.8 (351.01)

8. Primary Outcome: Pharmacokinetic: Cmax of Betamethasone 17-propionate
Description: The mean Cmax (Maximum Observed Plasma Concentration) of betamethasone 17- propionate was determined
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | 101.5 (77.551)

9. Primary Outcome: Pharmacokinetic: Cmax of Betamethasone 17-propionate
Description: The mean Cmax (Maximum Observed Plasma Concentration) of betamethasone 17- propionate was determined
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | 116 (64.826)

10. Primary Outcome: Pharmacokinetic: AUClast of Betamethasone 17-propionate
Description: The mean AUClast (Area under the Plasma Concentration-Time Curve from Time 0 to the Last Observed Measurable Concentration) for betamethasone 17-propionate was determined
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | 1036.7 (1885.01)

11. Primary Outcome: Pharmacokinetic: AUClast of Betamethasone 17-propionate
Description: as for outcome 10
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | 570.92 (517.107)

12. Primary Outcome: Pharmacokinetic: AUClast of Betamethasone 17-propionate
Description: as for outcome 10
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | 634.65 (467.426)

13. Primary Outcome: Pharmacokinetic: Cmax of Calcipotriol
Description: The mean Cmax (Maximum Observed Plasma Concentration) of calcipotriol was determined
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | 107.6 (NA) — The pharmacokinetic parameter could not be reliably estimated

14. Primary Outcome: Pharmacokinetic: Cmax of Calcipotriol
Description: The mean Cmax (Maximum Observed Plasma Concentration) of calcipotriol was determined
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

15. Primary Outcome: Pharmacokinetic: Cmax of Calcipotriol
Description: The mean Cmax (Maximum Observed Plasma Concentration) of calcipotriol was determined
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

16. Primary Outcome: Pharmacokinetic: AUClast of Calcipotriol
Description: The mean AUClast (Area under the Plasma Concentration-Time Curve from Time 0 to the Last Observed Measurable Concentration) for calcipotriol was determined
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | 169.6 (NA) — The pharmacokinetic parameter could not be reliably estimated

17. Primary Outcome: Pharmacokinetic: AUClast of Calcipotriol
Description: as for outcome 16
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

18. Primary Outcome: Pharmacokinetic: AUClast of Calcipotriol
Description: as for outcome 16
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

19. Primary Outcome: Pharmacokinetic: Cmax of MC1080
Description: The mean Cmax (Maximum Observed Plasma Concentration) of MC1080 was determined
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | 95.35 (NA) — The pharmacokinetic parameter could not be reliably estimated

20. Primary Outcome: Pharmacokinetic: Cmax of MC1080
Description: The mean Cmax (Maximum Observed Plasma Concentration) of MC1080 was determined
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | 57.57 (36.218)

21. Primary Outcome: Pharmacokinetic: Cmax of MC1080
Description: The mean Cmax (Maximum Observed Plasma Concentration) of MC1080 was determined
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

22. Primary Outcome: Pharmacokinetic: AUClast of MC1080
Description: The mean AUClast (Area under the Plasma Concentration-Time Curve from Time 0 to the Last Observed Measurable Concentration) for MC 1080 was determined
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | 430.9 (NA) — The pharmacokinetic parameter could not be reliably estimated

23. Primary Outcome: Pharmacokinetic: AUClast of MC1080.
Description: To assess the The mean AUClast (Area under the Plasma Concentration-Time Curve from Time 0 to the Last Observed Measurable Concentration) for MC 1080 was determined
Time Frame: Day 7
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | 221.2 (175.16)

24. Primary Outcome: Pharmacokinetic: AUClast of MC1080.
Description: as for outcome 22
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
h*pg/mL | NA (NA) — The pharmacokinetic parameter could not be reliably estimated

25. Secondary Outcome: Efficacy: Percentage Change in m-PASI From Baseline to Day 28
Description: Psoriasis Area and Severity Index (PASI) is based on the investigator's assessment of the disease.
  The extent and severity of redness, thickness and scaliness of psoriasis are recorded for three regions (arms, trunk and legs) and these are used to calculate PASI. The PASI can range between 0 (best) to 64.8 (worst). m-PASI indicate that the scale is modified.
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
percentage of change | -72.4 (24.5)

26. Secondary Outcome: Efficacy: Subjects With 'Clear' or 'Almost Clear' Disease by Investigator's Global Assessment at Day 28.
Description: Subjects with 'clear' or 'almost clear' disease by investigator's globala ssessment at day 28.
  Investigator global assessment (IGA) is based on the investigator's assessment of the disease severity (Plaque thickening, Scaling and Erythema) using a 6-point scale (Clear,Almost clear, Mild,Moderate, Severe, and Very severe). The assessment represents the average lesion severity on the trunk and limbs. IGA can range between 1 (best) and 6 (worst). The assessment is based on the condition of the disease at the time of evaluation, and not in relation to the condition at a previous visit.
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | LEO 90105 Ointment
Number analyzed (Participants) | 13
participants | 6

ADVERSE EVENTS:
Arm/Group | LEO 90105 Ointment
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 90105 Ointment (N=13)
Abdominal discomfort (Gastrointestinal disorders) | 1
Folliculitis (Infections and infestations) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO acknowledges the investigators right to publish the entire results of the study, irrespective of outcome. LEO retains the right to have any publication submitted to LEO for review. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.